CLINICAL TRIAL: NCT02229019
Title: The Southampton Mealtime Assistance Roll-out Trial
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MED1203; 14/LO/1363 (Other: London-Chelsea Research Ethics Committee)
Record Dates: First submitted 2014-08-20; First posted 2014-08-29 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Volunteer Mealtime Assistants
Keywords: Volunteers; Mealtime assistance; Older adults; Nutrition; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volunteer mealtime assistance (Experimental): Trained volunteers will provide mealtime assistance to older hospital inpatients at one mealtime each weekday.
  Interventions: Behavioral: Volunteer mealtime assistance

INTERVENTIONS:
Behavioral: Volunteer mealtime assistance

SUMMARY:
The Southampton Mealtime Assistance Study aims to determine whether it is feasible and acceptable to introduce trained volunteers as mealtime assistants in five different departments of one large hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 70 years admitted to one of the wards under study

Exclusion Criteria:

* Patients with active bowel pathology
* Patients in the terminal phase of their life
* Patients who are artificially fed (parenterally or enterally)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of volunteer mealtime assistants in different hospital departments | 16 months
  Is it feasible to recruit and sustain sufficient volunteers to provide mealtime assistance across a large hospital trust? Are these volunteers acceptable to patients, relatives, and staff? This will be determined by recording the number of volunteers recruited, trained and assessed and by recording their activity, in numbers of mealtimes assisted per week and duration of volunteering. If a volunteer discontinues their role, the reasons will be identified for this.
  Acceptability will be assessed through qualitative methods- interviews with patients and relatives and focus groups with nursing staff and volunteers.

SECONDARY OUTCOMES:
Changes in food choice and dietary intake before and after the introduction of volunteer mealtime assistants | 16 months
  The food choices and dietary intake of patients on the wards under study will be determined twice prior to the introduction of the volunteers and twice after their introduction. This will take place at the mealtime where the volunteers are assisting. The weight of meals served is portion controlled by the hospital caterers to within 10% of the stated weight. Therefore, using these stated weights and by measuring the leftover weight of food, we will calculate each patient's dietary intake at that mealtime.
Costs to the hospital trust associated with implementing a volunteer mealtime assistance programme | 16 months
  Staff costs in terms of time spent training and supporting volunteers will be recorded, as will any consumables required for the study. The costs will be totalled to provide an overall cost estimate of implementing a volunteer mealtime assistance programme.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Rossiter, MBChB, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Howson FFA, Robinson SM, Lin SX, Orlando R, Cooper C, Sayer AAP, Roberts HC. Can trained volunteers improve the mealtime care of older hospital patients? An implementation study in one English hospital. BMJ Open. 2018 Aug 5;8(8):e022285. doi: 10.1136/bmjopen-2018-022285. PMID 30082361